CLINICAL TRIAL: NCT00336258
Title: US-Doppler and Procoagulant Microparticles for the Diagnosis of Asymptomatic DVT in Advanced Cancer Patients With Poor Performance Status
Status: Completed | Type: Observational
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Dr Beck-Razi N, Rambam medicl center
Other Study IDs: BECKCTIL
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2007-04

CONDITIONS: Deep Vein Thrombosis; Cancer
Keywords: Deep Vein Thrombosis; Cancer; US- Doppler; Procoagulant Microparticles; Asymptomatic
MeSH Terms: conditions — Venous Thrombosis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The aim of this study is to determine the prevalence of asymptomatic lower extremity DVT detected by US-Doppler and procoagulant microparticles in a selected group of cancer patients suffering from an advanced stage of the disease.

An attempt will be made to determine whether there is a correlation between this prevalence and various clinical and laboratory parameters.

DETAILED DESCRIPTION:
The association between malignancy and venous thromboembolism(VTE) is well known. VTE is one of the most common complications seen in cancer patients Early detection of VTE can identify patients who may benefit from anticoagulant therapy and prevent morbidity and mortality.

There are recommendations for hospitalized cancer patients who are bedridden with an acute medical illness to receive prophylaxis, but in practice this is not clear cut.It has been shown, in other selected groups of patients that Ultrasound Doppler can be used in order to diagnose asymptomatic DVT (deep vein thrombosis). Hematological coagulation tests, including procoagulant microparticles will be performed for the evaluation of coagulation profile, in order to evaluate the possible correlation between the prevalence of asymptomatic DVT and these laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients with an advanced stage of the disease, hospitalized in the oncology department.
* WHO performance status of 3( i.e. spends more than half his/her time in bed or seated) - or 4 ( i.e. completely confined to bed or to chair) : for at least a week; according to the treating physician, the poor performance status results from advanced malignancy.
* Patient is asymptomatic for lower extremity DVT according to the treating physician

Exclusion Criteria:

* major surgery during more than a month, from the time of investigation
* anticoagulant therapy for more than one month, from the time of investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with an advanced stage of the disease, hospitalized in the oncology department.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nira Beck-Razi, Principal Investigator — Ministry of Health, Israel
Locations (1):
- Rambam medical center, Haifa, Israel